CLINICAL TRIAL: NCT06431165
Title: Effects of Different Doses of Intravenous Lidocaine Infusion on Peri-operative Pain and Incidence of Postoperative Chronic Pain Within ERAS Protocols, a Dose Finding Study.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Yahia El Sayed Kamel, Lecturer of anesthesiology and surgical ICU and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pain management
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Perioperative Pain Management

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled double blinded study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each patient will be assigned by a randomly computer generated number to one of the 3 groups and the group assignment will be put in a sealed envelope only accessible by the investigator responsible for preparing the drug syringes. The patient and data collectors will be blinded to the patient group allocation as well as the managing anesthiologists during the operation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Group A: Bolus 10 ml Syringe with Lidocaine 0.5% (2.5 ml lidocaine 2% + 7.5 ml N.S), and infusion 50 ml Syringe with Lidocaine 0.5% (12.5 ml Lidocaine 2% + 37.5 ml N.S).
  Interventions: Drug: Lidocaine IV
- Group B (Active Comparator): Group B: Bolus 10 ml Syringe with Lidocaine 1% (5 ml lidocaine 2% + 5 ml N.S), and infusion 50 ml Syringe with Lidocaine 1% (25 ml Lidocaine 2% + 25 ml N.S).
  Interventions: Drug: Lidocaine IV
- Group C (Active Comparator): Group C: Bolus 10 ml Syringe with plain Lidocaine 2%, and infusion 50 ml Syringe with plain Lidocaine 2%.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — After confirming patient history, type of operation and patient group allocation, standard ASA monitoring will be attached to the patient then the I.V induction of anesthesia will be commenced using standard doses of Propofol &Tracrium in addition to 1 μg/kg Fentanyl and 1 ml/10 kg from the bolus Lidocaine syringe followed after 3 minutes by endotracheal intubation, then the Lidocaine infusion Syringe will be attached to a separate I.V line at an infusion rate of 1 ml/10 kg/h. The patient will receive 1 gm of I.V paracetamol and the surgery will be allowed to proceed.

SUMMARY:
This study aimed To investigate the effects of different doses of Intraoperative intravenous lidocaine infusion on intraoperative opioid consumption, perioperative pain control and incidence of postoperative chronic pain.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) protocols or fast track surgery are a number of interventions which are carried out in the perioperative period. They are aimed to decrease the harmful effects of surgery on the body and help the patient recover better after surgery. ERAS has been shown to reduce the length of hospital stay, overall hospital costs, opioid consumption in the perioperative period and to reduce complication rates.

One of the most important components of ERAS is adequate perioperative pain control using a multi-modal analgesic approach to help decrease dependence on opioids and provide better recovery and less postoperative hospital stay. Also, the severity and duration of acute postoperative pain is one of the predictors of chronic postsurgical pain (CPSP). Neuroplasticity (spinal sensitization) following the trauma of surgery can transform an acute pain to chronic pain if not treated effectively by aggressive management of acute pain.

Lidocaine (or 2-(diethylamino)-N-(2.6-dimethylphenyl) acetamide) is the main prototype of amino-amide local anesthetics. It has analgesic, anti-hyperalgesic and anti-inflammatory properties, which enable its use as a general anesthetic adjuvant. It can reduce nociception, cardiovascular responses to surgical stress, postoperative pain, and analgesic requirements.

Accordingly, Lidocaine infusion can have a role in enhancing postoperative quality of recovery, decreasing incidence of chronic postoperative pain and even increasing overall survival in patients undergoing major surgeries like in pancreatectomy.

The Systemic effects of intravenous Lidocaine infusion depends on its plasma level which is affected by the rate and dose of administration, drug interactions and speed of metabolism and elimination. Around 90% of lidocaine undergoes hepatic metabolism (CYP3A4), with the production of active metabolites. During lidocaine continuous infusion, the accumulation of these metabolites may inhibit its biotransformation and might be involved in some cases of intoxication. The clearance rate of lidocaine is approximately 0.85 L/kg/h. Finally, lidocaine is eliminated by the kidney (10% of lidocaine is eliminated unchanged in the urine).

The target plasma concentrations for Lidocaine for providing effective analgesia is 2.4 ± 0.6 μg/mL, while side effects as - have been reported when the plasma concentration was higher than 5-8 μg/mL. The suggested dosing regimens mentioned in literature to achieve this effective plasma level while avoiding toxicity is a bolus of 1-2 mg/kg at surgery start followed by infusion of 1-2 mg/kg/h over the duration of the surgery which is a relatively wide range, specially, considering the wide variability in type and duration of surgeries, demographics, physical and medical status of patients and type of anesthetic agents and drugs used which all can affect Lidocaine activity, elimination & toxicity.

To the best of our knowledge, no evidence exist in the literature that can point towards the ideal dosing regimen for intravenous Lidocaine infusion that can achieve the desired valuable clinical effects while decreasing the incidence of adverse side effects among the wide variety of surgeries and patients encountered within ERAS protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 65.
* Patients with ASA I and II status.
* Patients undergoing open laparotomy surgeries (including open cholecystectomies).

Exclusion Criteria:

* Patients unable to comprehend the informed consent.
* Patients on long term pre-operative opioid regimens.
* Patients with impairment in hepatic or renal functions.
* Patients who are planned to receive any form of regional block for the surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Total Intraoperative opioid consumption (Fentanyl) | Every five minutes
  Fentanyl doses of 0.5 mic/kg will be given when there is increase in hemodynamics by 20% of baseline and this will be reported

SECONDARY OUTCOMES:
Total opioid consumption (Morphine) in the first 24 hours postoperative. | Every one hour postoperative for 24 hours
Time of first rescue analgesia used in the first 24 hours postoperative | Every one hour postoperative for 24 hours
  Time between end of surgery and the first dose of rescue analgesia administered to the patient
Incidence of side effects related to Lidocaine infusion during the first 24 hours postoperative. | Every one hour postoperative for 24 hours
Incidence of chronic postoperative pain 2 months after the surgery. | Every week for 2 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ahmed Mansour, Assistant professor, Study Director — Cairo University; Islam Ayman Mohammed Shawky, MD, Study Director — Cairo University; Nora Amr Agiza, MD, Study Director — Cairo University; Omnia Y Kamel, MD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No